CLINICAL TRIAL: NCT03355547
Title: Observation of Atelectasis Using Lung Ultrasonography in Children Undergoing General Anesthesia: the Cohort Study for Evaluation of the Relationship Between the Incidence and Severity of Upper Respiratory Tract Infection and the Magnitude of Anesthesia-induced Atelectasis
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0766
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- no URI (upper respiratory tract infection) symptoms: Patients without upper respiratory tract infection symptoms
  Interventions: Other: questionnaire about the severity of their symptoms of upper respiratory tract infection
- URI (upper respiratory tract infection) symptoms: Patients with upper respiratory tract infection symptoms
  Interventions: Other: questionnaire about the severity of their symptoms of upper respiratory tract infection

INTERVENTIONS:
Other: questionnaire about the severity of their symptoms of upper respiratory tract infection — Before the operation, the researcher interviews the parents of the pediatric patients to check whether they have the upper respiratory tract infection and asks them to fill out a questionnaire about the severity of their symptoms. The questionnaire consists of 8 types of symptom about upper respiratory infections and each symptom was checked from 0 to 3 according to severity by their patients.

SUMMARY:
Pediatric patients between 6months and 6years old will be included. They are scheduled for elective general or urologic surgery at a single tertiary medical center. Before the operation, the researcher interviews the parents of the pediatric patients to check whether they have the upper respiratory tract infection and asks them to fill out a questionnaire about the severity of their symptoms. The researcher will get the symptom score of the upper respiratory tract infection in the questionnaire. The degree of anesthesia induced atelectasis is measured using lung ultrasound. Pulmonary ultrasound is performed after endotracheal intubation and at the end of the operation dividing the patient's thorax into 12 regions. The investigator grades the degree of atelectasis at each region form 0 to 3 points. After the end of the operation, check whether the respiratory adverse effects occurred during emergence and recovery at the post anesthesia care unit.

ELIGIBILITY:
Inclusion Criteria:

* Age: Pediatric patients older than 6 months and younger than 6 years
* scheduled for elective pediatric general or urology surgery.

Exclusion Criteria:

* undergoing laparoscopic surgery
* pediatric patients with lower respiratory tract infection( pneumonia , bronchiolitis )
* patients with bronchopulmonary dysplasia history
* hemodynamic instability

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients between 6months and 6years old scheduled for elective general or urologic surgery at a single thetiary medical center.
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
The degree of atelectasis due to general anesthesia using lung ultrasound | The investigator will measure the degree of atelectasis using lung ultrasound at 2 minutes after endotracheal intubation and at 5minutes the end of the operation.
  Anesthesia induced atelectasis is diagnosed when the ultrasound findings as B-line (appears hyperechoic lines perpendicular to the pleura) and consolidation(loss of pleural line and hypoechoic area) are identified. The chest is divided into 12 regions: three longitudinal lines (parasternal, anterior, and posterior axillary) and two axial lines (above the diaphragm, and 1cm above the nipples) in each hemithorax. The investigator grades the degree of atelectasis at each region form 0 to 3 points. The degree of juxtapleural consolidation was graded: (a0) no consolidation; (a1) minimal juxtapleural consolidation; (a2) small-sized consolidation(<50%); and (a3) large-sized consolidation(>50%). The degree of B-lines was divided into four grades: (b0) fewer than three isolated B-lines; (b1) multiple well-deﬁned B-lines; (b2) multiple coalescent B-lines; and (b3) white lung.

SECONDARY OUTCOMES:
Occurrence of respiratory adverse effects after the operation | 10 minutes after extubation at the post anesthesia care unit
  After the end of the operation, check whether the respiratory adverse effects occurred when the patient is extubated and 10, 30 minutes after extubation at the post anesthesia care unit. Respiratory adverse effects are bronchospasm and laryngospasm. We analyze the symptom score of upper respiratory tract infection in pediatric patients who showed respiratory adverse events and suggest the cut off value of the score with high risk of respiratory adverse events by multivariate logistic regression.
Occurrence of respiratory adverse effects after the operation | 30 minutes after extubation at the post anesthesia care unit
  After the end of the operation, check whether the respiratory adverse effects occurred when the patient is extubated and 10, 30 minutes after extubation at the post anesthesia care unit. Respiratory adverse effects are bronchospasm and laryngospasm. We analyze the symptom score of upper respiratory tract infection in pediatric patients who showed respiratory adverse events and suggest the cut off value of the score with high risk of respiratory adverse events by multivariate logistic regression.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine Anesthesia and Pain Research Institute Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee HM, Byon HJ, Kim N, Gleich SJ, Flick RP, Lee JR. Effect of upper respiratory infection on anaesthesia induced atelectasis in paediatric patients. Sci Rep. 2021 Mar 16;11(1):5981. doi: 10.1038/s41598-021-85378-0. PMID 33727626